CLINICAL TRIAL: NCT05785286
Title: To Linguistically and Psychometrically Validate the Hong Kong Chinese Version of the BPH 3-item Questionnaire.
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2022.645
Record Dates: First submitted 2023-02-27; First posted 2023-03-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subject with male LUTS: Male subjects who have been bothered by male LUTS for at least 4 weeks and are still able to pass urine on their own without the need of assistance or urethral catheterization.
  Interventions: Other: BPH 3-item questionnaire
- Subject who is waiting for their transurethral ablative prostate surgery: Male subjects who are waiting for BPH surgery and are still able to pass urine on their own without the need of assistance or urethral catheterization.
  Interventions: Other: BPH 3-item questionnaire

INTERVENTIONS:
Other: BPH 3-item questionnaire — BPH 3-item questionnaire. The questionnaire consists of only three items. A raw score ranging from 0 to 5 is assigned to each of the items, giving a final total score varying from 0 (no symptom) to 15 (very symptomatic).

SUMMARY:
This study is to linguistically and psychometrically validate the translated and culturally adapted Hong Kong Chinese version of the BPH 3-item questionnaire.

DETAILED DESCRIPTION:
A new BPH 3-item questionnaire has recently been developed and published, and it may serve as a screening tool for male-LUTS due to symptomatic BPE. The questionnaire consists of only three items. A raw score ranging from 0 to 5 is assigned to each of the items, giving a final total score varying from 0 (no symptom) to 15 (very symptomatic). This questionnaire has been translated and validated into five different European languages and was harmonized cross-culturally for linguistic validation, followed by psychometric accuracy testing.

This new questionnaire may help rationalize more early commencement of therapy aimed at reducing the prostate size for the treatment of male LUTS due to BPE.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 90 years old Chinese male subjects presented with male-LUTS for at least 4 weeks
* The subjects are able to read and fully comprehend with the content of the questionnaires
* The subjects are willing to give informed consent for the study

Exclusion Criteria:

* peak uroflow ≤4mL/sec;
* post-void residual (PVR) ≥300 mL;
* unable to give informed consent
* need of clean intermittent self-catheterization / indwelling urethral catheterization at the time of enrolment;
* Surgical treatment (e.g. TURP) of bladder outlet obstruction / symptomatic benign prostate enlargement (BPE) ≤ 3 months before entry into the study
* clinical suspicion / presence of untreated urethral stricture and/or bladder neck stenosis,
* clinical suspicion / presence of genitourinary cancer including active prostate cancer with ongoing surgical or radiation treatment, or the need of treatment, or bladder cancer, or persistent unexplained hematuria;
* uncontrolled heart failure / diabetes mellitus(DM) / hypertension(HT);
* neuropathic bladder;
* Currently on dialysis or in consideration for dialysis due to end stage renal disease;
* More than 3 urinary tract infections within the last 12 months;
* Unstable dose of diuretic within the past 3 months;
* Has an artificial urinary sphincter;
* Impaired mental status;
* male-LUTS due to urinary tract infections / chronic prostatitis / chronic pelvic pain

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Male subjects who have been bothered by male LUTS for at least 4 weeks and are still able to pass urine on their own without the need of assistance or urethral catheterization at the time of enrolment. Or male-LUTS subject who is waiting for their transurethral ablative prostate surgery for their symptomatic BPE.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Reliability of BPH 3-item questionnaire | up to 24 weeks
  Reliability was assessed by internal consistency and test-retest correlation. (ρ) correlation, with the IPSS (total score / voiding domain (ie Q.1, 3, 5, 6) and prostate volume measured by TRUS.
Internal consistency of BPH 3-item questionnaire | up to 24 weeks
  Internal consistency was assessed by Cronbach's alpha coefficients, with >0.7 being considered acceptable
Test-retest reliability of BPH 3-item questionnaire | up to 24 weeks
  Test-retest reliability was assessed by intra-class correlation coefficient. Values between 0.6 and 0.8 indicate substantial agreement, and values over 0.8 indicate near-perfect agreement
The convergent validity of the BPH 3-item questionnaire | up to 24 weeks
  was estimated by Spearman rho (ρ) correlation, with the IPSS (total score / voiding domain (ie Q.1, 3, 5, 6) and prostate volume measured by TRUS.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Alice Ho Miu Ling Nethersole Hospital, Hong Kong
  - Prince of Wales Hospital, Shatin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu PSK, Leung CLH, Cheung MH, Woo SWS, Lo TK, Chan TNH, Wong WKK. Hong Kong Geriatrics Society and Hong Kong Urological Association consensus on personalised management of male lower urinary tract symptoms in the era of multiple co-morbidities and polypharmacy. Hong Kong Med J. 2021 Apr;27(2):127-139. doi: 10.12809/hkmj209049. PMID 33879628
- [Background] Tubaro A, Niero M, Adalig B, Lulic Z, Plastino J, Kimbrough C, Manyak MJ. Evaluation of a 3-item screening tool to identify men with benign prostatic enlargement/obstruction in a primary care cohort. Minerva Urol Nephrol. 2022 Feb;74(1):85-92. doi: 10.23736/S2724-6051.20.03834-5. Epub 2020 Sep 29. PMID 32993275
- [Background] Chiu PK, Ng CF, Semjonow A, Zhu Y, Vincendeau S, Houlgatte A, Lazzeri M, Guazzoni G, Stephan C, Haese A, Bruijne I, Teoh JY, Leung CH, Casale P, Chiang CH, Tan LG, Chiong E, Huang CY, Wu HC, Nieboer D, Ye DW, Bangma CH, Roobol MJ. A Multicentre Evaluation of the Role of the Prostate Health Index (PHI) in Regions with Differing Prevalence of Prostate Cancer: Adjustment of PHI Reference Ranges is Needed for European and Asian Settings. Eur Urol. 2019 Apr;75(4):558-561. doi: 10.1016/j.eururo.2018.10.047. Epub 2018 Nov 2. PMID 30396635
- [Background] Stravodimos KG, Petrolekas A, Kapetanakis T, Vourekas S, Koritsiadis G, Adamakis I, Mitropoulos D, Constantinides C. TRUS versus transabdominal ultrasound as a predictor of enucleated adenoma weight in patients with BPH: a tool for standard preoperative work-up? Int Urol Nephrol. 2009 Dec;41(4):767-71. doi: 10.1007/s11255-009-9554-9. Epub 2009 Apr 7. PMID 19350408